CLINICAL TRIAL: NCT05828303
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Potential Drug Interactions Between Repotrectinib and Metformin, Digoxin, and Rosuvastatin in Patients With Advanced Solid Tumors Harboring ROS1 or NTRK1-3 Rearrangements
Brief Title: A Phase 1 Study to Evaluate the Potential Drug Interactions Between Repotrectinib and Metformin, Digoxin, and Rosuvastatin in Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1027
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2023-03-28; First posted 2023-04-25 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — repotrectinib; Metformin; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Repotrectinib (TPX-0005) (Experimental): Phase 1 Oral repotrectinib (TPX-0005) + cocktail drugs (metformin hydrochloride, digoxin, rosuvastatin calcium)
  Interventions: Drug: TPX-0005; Drug: Metformin Hydrochloride; Drug: Digoxin; Drug: Rosuvastatin Calcium

INTERVENTIONS:
Drug: TPX-0005 — Oral TPX-0005 capsules
  Other Names: repotrectinib
Drug: Metformin Hydrochloride — oral solution
  Other Names: Glucophage; Metabet; Glucient; Diagemet; Axpinet
Drug: Digoxin — oral tablet
  Other Names: Lanoxin
Drug: Rosuvastatin Calcium — oral tablet
  Other Names: Crestor

SUMMARY:
This is a Phase 1 study to evaluate the potential drug-drug interaction (DDI) effect of repotrectinib on certain drug transporters in patients with advanced cancer.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, fixed-sequence study to evaluate the potential drug-drug interaction (DDI) effect of repotrectinib on drug transporters (metformin, digoxin and rosuvastatin) following multiple dose administration of repotrectinib in patients with advanced cancer harboring ROS1 and NTRK1 Rearrangements.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of locally advanced, or metastatic solid tumor (including primary central nervous system [CNS] tumors) that harbors a ROS1 or NTRK1-3 gene fusion.
2. Patient must have a documented ROS1 or NTRK1-3 gene fusion determined by tissue-based local testing.
3. Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 (≥ 18 years).
4. Protocol specified baseline hematology, liver function and kidney function laboratory values.

Key Exclusion Criteria:

1. Concurrent participation in another therapeutic clinical trial.
2. Symptomatic brain metastases or leptomeningeal involvement.
3. Major surgery within 4 weeks of start of repotrectinib treatment.
4. Clinically significant cardiovascular disease.
5. History of non-pharmacologically induced prolonged QTc interval
6. Known active infections requiring ongoing treatment (bacterial, fungal, viral including human immunodeficiency virus positivity).
7. Gastrointestinal disease or other malabsorption syndromes.
8. Current or anticipated use of drugs that are known to be moderate or strong CYP3A inhibitors or inducers.
9. Patients who have received, or are expected to receive metformin, digoxin or rosuvastatin within 14 days prior to beginning of the DDI assessment period.
10. Patients who have received or are expected to receive drugs that are inhibitors of P-gp, OATP1B1, BCRP, and MATE2-K within 14 days or 5 half-lives (whichever is longer) prior to beginning of the DDI assessment period until the DDI assessment period is completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Area under plasma-concentration time curve | Within 28 days of first cocktail dose
  AUC0-t: area under the plasma-concentration time curve from time 0 to time of the last measurable concentration. AUC0-inf: area under the plasma-concentration time curve from time 0 to infinity (if data permit).
Maximum Observed Plasma Concentration | Within 28 days of first cocktail dose
  Cmax: maximum observed plasma concentration

SECONDARY OUTCOMES:
Evaluate safety and tolerability | Within 28 days of first cocktail dose
  To evaluate the safety and tolerability of repotrectinib in patients with moderate and severe hepatic impairment and patients with normal hepatic function following single and multiple dose administration of repotrectinib assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (2):
  - Gabrail Cancer Research Center, Canton, Ohio
  - Local Institution - 2101, Canton, Ohio
- Local Institution - 2119, Westmead, New South Wales, Australia
- Brazil (5):
  - Local Institution - 2126, Botafogo, Rio de Janeiro
  - Local Institution - 2132, Porto Alegre, Rio Grande do Sul
  - Local Institution - 2134, Porto Alegre, Rio Grande do Sul
  - Local Institution - 2130, São Paulo, São Paulo
  - Local Institution - 2108, São Paulo
- France (7):
  - Local Institution - 2123, Bordeaux
  - Local Institution - 2122, La Tronche
  - Local Institution - 2117, Marseille
  - Local Institution - 2115, Nantes
  - Local Institution - 2121, Poitiers
  - Local Institution - 2136, Rennes
  - Local Institution - 2120, Saint-Herblain
- Italy (6):
  - Local Institution - 2135, Milan, MI
  - Local Institution - 2116, Rozzano, MI
  - Local Institution - 2111, Perugia, PG
  - Local Institution - 2104, Aviano, PN
  - Local Institution - 2103, Verona, VR
  - Local Institution - 2114, Naples
- Spain (12):
  - Local Institution - 2124, Barcelona, B
  - Local Institution - 2113, Barcelona, B
  - Local Institution - 2105, Barcelona, B
  - Local Institution - 2129, Pozuelo de Alarcón, Madrid
  - Local Institution - 2138, Madrid, M
  - Local Institution - 2110, Madrid, M
  - Local Institution - 2128, Madrid, M
  - Local Institution - 2109, Barcelona
  - Local Institution - 2127, Madrid
  - Local Institution - 2106, Madrid
  - Local Institution - 2112, Pamplona
  - Local Institution - 2125, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com